CLINICAL TRIAL: NCT03351712
Title: ACTonHEALTH Study Protocol: Promoting Psychological Flexibility With Activity Tracker and mHealth Tools to Foster Healthy Lifestyle for Obesity and Other Chronic Health Conditions
Brief Title: mACTonHEALTH: Psychological Flexibility and Activity Tracker - Protocol
Acronym: ACTonHEALTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 03C701
Record Dates: First submitted 2017-11-07; First posted 2017-11-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Health Behavior
Keywords: Wearables; Activity Trackers; ACT; Health promotion; Obesity; Chronic Health Condition; Psychological well-being; Quality of life; Behavior modification; RCT
MeSH Terms: conditions — Health Behavior; Obesity; Psychological Well-Being | interventions — Fitness Trackers

STUDY DESIGN:
Intervention Model Description: Single subject design and group design combined
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gold Standard Intervention + Activity Tracker WITHOUT Feedback (Active Comparator): Gold Standard Intervention + Activity Tracker WITHOUT Feedback (Medical Rehabilitation, Motivational Support and Psycho-Education) During the in-patient phase, participants will participate in the intensive four-week hospital-based and medically-managed rehabilitation program for weight reduction. All patients will be placed on a hypocaloric nutritionally balanced diet tailored to the individual after consultation with a dietitian. Furthermore, they will receive nutritional counseling provided by dietitians, have physical activity training provided by physiotherapists and motivational support with elements of psycho-education provided by physicians trained and informed by psychologists-psychotherapists.
  Interventions: Behavioral: Gold Standard Intervention + Activity Tracker WITHOUT Feedback
- Gold Standard Intervention and Activity Tracker WITH Feedback (Experimental): In this experimental condition, will be provided the same rehabilitation program for the 4-weeks in-patient phase. In addition, for these subjects will be implemented a Stepped Protocol using wearable devices / activity trackers to collect information about daily physical activity and providing meaningful and informative feedbacks. The additional procedure starts during the in-patients phase, delivering and explaining the use of the wearable devices. In this meeting, longer than the one previously described for the control condition, experimenters provide information, set individualized goals and explain feedbacks which will be delivered after ending in-patients phase by the electronic wearable devices.
  Interventions: Behavioral: Gold Standard Intervention and Activity Tracker WITH Feedback
- ACT-Based Intervention and Activity Tracker WITHOUT Feedback (Experimental): In this experimental condition, the subjects followed the normal medical rehabilitation program described above for the first experimental condition. For the out-patient phase the ACT intervention includes monthly 30 minutes skype-telephone sessions. The ACT-based interventions includes different processes: 1) Acceptance, that involves the active awareness of difficult private experiences without attempts to control or avoid unpleasant emotions. 2) Mindfulness, refers to engaging in present moment experience and adopting an open and curious attitude. 3) Defusion: Participants will be encouraged to defuse from thoughts and feelings by turning attention toward the 'noticing-self', instead of becoming attached to thoughts and 'run' through life on 'auto-pilot'. 4) Values and Commitment: encouraging participants to live in accordance with their values, participants can engage in meaningful activities despite experiencing unwanted emotions/ sensations.
  Interventions: Behavioral: ACT-Based Intervention and Activity Tracker WITHOUT Feedback
- ACT-Based Intervention and Activity Tracker WITH Feedback (Experimental): ACT-Based Intervention and Activity Tracker WITH Feedback (Combining ACT and Behavioral Change) In the last experimental condition, obese individuals will follow the same rehabilitation program in the in-patients phase of the Behavioral Change condition, with the addition of the brief ACT intervention of 4 45-minutes sessions for a total amount of 3 hours one-to-one therapy sessions, exactly as in the ACT condition. In the out-patient phase of 16 weeks, each participant receive feedback from activity tracker following the same stepped protocol but message and feedbacks are informed by ACT therapist, including Value-based goal setting, prompt for including defusion from difficult thoughts, mindfulness cues and a set of ACT-consistent metaphors and messages.
  Interventions: Behavioral: ACT-Based Intervention and Activity Tracker WITH Feedback

INTERVENTIONS:
Behavioral: ACT-Based Intervention and Activity Tracker WITH Feedback — Combining ACT and Behavioral Change
  Arms: ACT-Based Intervention and Activity Tracker WITH Feedback
Behavioral: Gold Standard Intervention + Activity Tracker WITHOUT Feedback — Medical Rehabilitation, Motivational Support and Psycho-Education
  Arms: Gold Standard Intervention + Activity Tracker WITHOUT Feedback
Behavioral: Gold Standard Intervention and Activity Tracker WITH Feedback — Behavioral Change Condition - Activity Tracker
  Arms: Gold Standard Intervention and Activity Tracker WITH Feedback
Behavioral: ACT-Based Intervention and Activity Tracker WITHOUT Feedback — ACT-Based Intervention Standalone
  Arms: ACT-Based Intervention and Activity Tracker WITHOUT Feedback

SUMMARY:
Obesity and overweight are growing steadily and becoming a global epidemic. Recent researches report a 64% of the adult population as overweight. The social and economical impact is increasing and the most of the rehabilitation programs, while effective in the short term, do not produce long lasting results. From a behavioral perspective an explanatory model can describe the phenomena with the lack of sources of reinforcement related to healthy habits in the daily-life context. The goal of this project, combining Acceptance and Commitment Therapy and Wearable Technology, is to develop an effective intervention, efficient and sustainable, which continues after ending of the hospitalization, providing adequate contingencies of reinforcement in the natural environment, integrating systematic measurements, continuous feedbacks and individualized, values-based objectives. Related goal-setting show a shift from results linked with weight loss towards action connected with healthy life-style.

DETAILED DESCRIPTION:
Background The condition of being overweight is an increasing problem worldwide, becoming an epidemic both in Europe and in the United States. Recent estimates that over 60% of adults are overweight and at the same time obesity affects around 35% of the population. In the US the cost of the health system to cope with obesity and related diseases now exceeds the sum of 100 billion and in Europe costs are currently similar. Health risks related to being overweight include psychological difficulties, depression and stigma, physical problems and heart diseases, cancer and respiratory diseases not to mention musculoskeletal and metabolic problems.

Obesity is a chronic health condition, but is also a major risk factor for various diseases both chronic and acute. This problem is currently steadily rising, with prevalence data and epidemiological estimates that should be of great concern. Despite strong biological components and hereditary aspects, obesity is primarily linked to incorrect habits of everyday life, mainly eating habits and physical activity. Numerous studies have documented that regular physical activity and wise choices in food uptake can prevent obesity and related conditions.

The main challenge in addressing obesity and associated disorders is represented by developing and making available and sustainable comprehensive programs that include combinations of physical activity, dietary aspects and psychological interventions.

Interventions developed in this way, including dietary education protocols, physical rehabilitation and exercises programs, nutritional, endocrinological, psychological, surgical and pharmacological treatments are mainly effective in the short term, despite many of which are characterized by high costs and several periods of hospitalization. The analysis of the literature suggests the superiority of intensive multidisciplinary interventions: health protocols, dietary programs, psychological and physical rehabilitation. One of the problems of such interventions is that they are often only possible during an hospitalization period, with high costs associated. However, despite good evidence of effectiveness, the long-term results are generally limited.

In general, availability, costs, compliance and long-term efficacy are important limitations to this variety of approaches. Frequently obese individuals regain about 30% of the weight they lost within the first year. After only 3 years they are returning to pre-treatment weight. Psychological intervention are generally assumed to be one of the core parts in the treatment aimed to obesity. In particular, Cognitive-Behavioral interventions, usually within multidisciplinary paths and rarely implemented individually, are generally considered the gold-standard for addressing the epidemic of obesity, or "globesity".

Rationale Reasons for the long-term failure of interventions for obesity can be found in the lack of long-term sources of reinforcement for healthy habits acquired during the intensive treatment period. The tradition of behavioral sciences has developed models of interpretation, explanation and pragmatic operation supported by evidence of effectiveness and efficiency in the promotion of desired behaviors in various contexts and with a longer time effect. These span from the cessation of smoking, passing trough the ability to adapt and live with chronic diseases, ending with the promotion of safety behaviors in working environments. For this reason behavior analysis in general, and in particular the Contextual Behavioral Science, can play a decisive role in the prevention of obesity and keeping the results achieved within short intensive protocols, usually held in hospitals.

By modifying deeply rooted and long-term acquired habits, the person with obesity can obtain more psychological and physical health, reduce risk factors and improve his overall health, wellness and quality of life with benefits not only for the individual but also for his social environment.

During the rehabilitation periods patients affected by obesity are frequently in contact with contingencies that are very different from those of their daily lives. In the rehabilitation facility or during the hospitalization, contingencies are efficiently shaped to promote desired behaviors and decrease actions that are identified as dysfunctional, with both aversive and reinforcing contingencies. Later on, after the treatment, in his natural environment initially behaviors are maintained, but having been promoted in a environment that provide contingencies supporting healthy behaviors, they often undergo a processes of extinction consequently with cessation of reinforce. At the same time, outside the hospital, dysfunctional behaviors such as avoiding physical activity and eating tasty food, are reinforced in a systematic and contingent way. This tendency to extinction of functional and healthy habits and reinforcement of dysfunctional habits leads, in the long term to gain the weight lost laboriously and this also leads to lower levels of well-being.

Although the existing programs already provide protocol phases to be implemented once they are home, often the patients fail to adhere to nutrition programs and planned activities. On the contrary they return frequently to previous habits, and show a high drop-out rate at follow-ups.

To overcome the limited long-term adherence after the hospitalization period, it is necessary to find a way to give significant, contingent and informative feedback also after the rehabilitation phase. In this regard the use of activity trackers represents a clear, valid and "smart" use of new technologies, linked to well established behavioral science.

Hypothesis, goals and expected results The project aims to promote a long-term change in lifestyle of as part of a multidisciplinary intervention, in close collaboration with physicians, the service of Clinical Nutrition and the osteo-articular rehabilitation.

The main goal of this study is test the efficacy of combining behavioral change technologies through contingent and meaningful feedbacks provided by wearable devices with ACT-based intervention, a well-studied psychological treatment developed in a contextual behavioral framework. The combination of thisapproach should be feasible and efficient, compared with gold standard treatment with inferior costs. Four experimental condition are provided: 1) usual care during hospitalization with programmed follow-up checks, 2) contingent feedback on daily life activities through activity trackers or wearable device stand-alone, 3) ACT based intervention stand-alone, 4). combination of the previous two, ACT-Based Intervention and Activity Tracker with Feedback.

Primary outcome, or dependent variable, of the study is physical activity as collected by wearable electronic devices. Other outcomes, as for example time of sleep, are collected by wearables, and other provided by self report through web platform. The independent variable of the study is the type of treatment (ACT intervention and feedbacks provided by activity trackers). For the purpose of the study we collect data about daily steps and workout log for each participants.

The intervention aims to help people in their everyday environment to remain more consistent with the choices made, and follow appropriate diets and physical activity. The project is directed to participants in the multidisciplinary rehabilitation program at St. Joseph Hospital - Verbania, Italian Auxological Institute, a private research institute that works also for the Italian national health system. The recruitment will take place progressively and subjects will be randomized to the four experimental conditions expected by the protocol. Data will be analyzed in different experimental single-subjects over multiple baselines designs. The subjects are also grouped according to the experimental condition to allow statistical analysis of experimental designs intergroup, consistent with the approach of a controlled and randomized trial.

Due to the novelty of using a combination of behavioral change strategies with Acceptance and Mindfulness - based therapy with wearable device to promote healthy life-style in the post-rehabilitation period, no well defined hypothesis have been established about the possible contribution of this kind of intervention in comparison with usual care, the "gold standard" multi-disciplinary treatment chronic conditions linked to obesity. With the development of mobile technology and brief clinical protocols, new interventions in the field of obesity and connected chronic pathologies have to be evaluated.

Anyway, the mACTonHEALTH study is quite innovative for different reasons. First, combination of single case designs with RCT is uncommon, particularly with medium-scale studies like this. Second, using wearable device activity trackers both as device for data collection measuring the primary outcomes and as device to provide contingent feedbacks, assumed to as one the two independent variable. Third, combining directly brief ACT intervention and behavior modification strategies with mobile-tech implementation is another element of innovation. Furthermore, although ACT is becoming well-studied in the traditional clinical context, large-scale application to both medical and natural settings has not largely occurred. Including in assessment procedure direct collectable data, indicators of both physical and psychosocial health. Also, the inclusion of objective physiological outcome measures constitutes an aspect of innovation in ACT research. Last, the study will focus on mediation mechanisms underlying treatment success and presents possible links to systematic models on psychological flexibility, a core process assessed in ACT researches.

Hypothesis To the best of the researcher's knowledge, this study will be the first randomized controlled trial to examine the effectiveness of a combination of contingent feedbacks provided with wearable devices with ACT-based interventions to improve healthy life style according to medical and behavioral prescription among obese patients. It is also one of the first example of a large implementation of multiple single case designs with a continuous data collection, made possible due the implementation of wearable-technology. Conducted in the context of clinical practice, this trial will potentially offer empirical support to alternative interventions to improve radical long-time change in life habits and consequently promote quality of life reducing mortality and morbidity rates among obese population. Furthermore, by virtue of its short duration, the program could potentially be utilized for health promotion also in non-hospitalization context and primary or secondary prevention of obesity and linked conditions.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years;
* obesity according to the WHO criteria (BMI ≥ 30); ù
* written and informed consent to participate, 4) tech-friendly to receive feedback through smartphone, mail and wearable devices

Exclusion Criteria:

* other severe psychiatric disturbance diagnosed by DSM-V criteria;
* severe visual difficulties,
* important limitations of movement, in particular subjects for which it is not recommended physical activity,
* concurrent medical condition not related to obesity. DSM-V (Thomas et al., 2014) will be used as screening tools for psychiatric disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity directly measured by wearable devices Daily STEPS Count | Baseline - after 4 weeks treatment - 6 months Follow Up - 12 months Follow Up - 18 months Follow Up -
  Daily Steps directly collected by wearable devices

SECONDARY OUTCOMES:
MDS - Mediterranean Diet Score | Baseline - after 4 weeks treatment - 6 months Follow Up - 12 months Follow Up - 18 months Follow Up -
  psychometric questionnaire about diet habits
PGWBI - Psychological General Well-Being Index | Baseline - after 4 weeks treatment - 6 months Follow Up - 12 months Follow Up - 18 months Follow Up -
  psychometric questionnaire assessing well-being
Acceptance & Action Questionnaire AAQ-II | Baseline - after 4 weeks treatment - 6 months Follow Up - 12 months Follow Up - 18 months Follow Up -
  psychometric questionnaire - a measure of Psychological Flexibility
International Physical Activity Questionnaires (IPAQ-SF) | Baseline - after 4 weeks treatment - 6 months Follow Up - 12 months Follow Up - 18 months Follow Up -
  Psychometric questionnaire that assesses Physical Activity

CONTACTS AND LOCATIONS:
Overall Officials: Gian Luca Castelnuovo, PhD, PsyD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- San Giuseppe Hospital, Istituto Auxologico Italiano IRCSS, Verbania, Italy

REFERENCES:
- [Background] Avena NM, Bocarsly ME, Hoebel BG, Gold MS. Overlaps in the nosology of substance abuse and overeating: the translational implications of "food addiction". Curr Drug Abuse Rev. 2011 Sep;4(3):133-9. doi: 10.2174/1874473711104030133. PMID 21999687
- [Background] Baranoff JA, Hanrahan SJ, Burke AL, Connor JP. Changes in Acceptance in a Low-Intensity, Group-Based Acceptance and Commitment Therapy (ACT) Chronic Pain Intervention. Int J Behav Med. 2016 Feb;23(1):30-8. doi: 10.1007/s12529-015-9496-9. PMID 26135404
- [Background] Behi R, Nolan M. Single-case experimental designs. 1: Using idiographic research. Br J Nurs. 1996 Nov 28-Dec 11;5(21):1334-7. doi: 10.12968/bjon.1996.5.21.1334. PMID 9015990
- [Background] Aldridge D. Single-case research designs for the clinician. J R Soc Med. 1991 May;84(5):249-52. doi: 10.1177/014107689108400502. No abstract available. PMID 2040997
- [Background] Bricker J, Wyszynski C, Comstock B, Heffner JL. Pilot randomized controlled trial of web-based acceptance and commitment therapy for smoking cessation. Nicotine Tob Res. 2013 Oct;15(10):1756-64. doi: 10.1093/ntr/ntt056. Epub 2013 May 23. PMID 23703730
- [Background] Byrne S, Cooper Z, Fairburn C. Weight maintenance and relapse in obesity: a qualitative study. Int J Obes Relat Metab Disord. 2003 Aug;27(8):955-62. doi: 10.1038/sj.ijo.0802305. PMID 12861237
- [Background] Carr KA, Daniel TO, Lin H, Epstein LH. Reinforcement pathology and obesity. Curr Drug Abuse Rev. 2011 Sep;4(3):190-6. doi: 10.2174/1874473711104030190. PMID 21999693
- [Background] Castelnuovo G, Manzoni GM, Pietrabissa G, Corti S, Giusti EM, Molinari E, Simpson S. Obesity and outpatient rehabilitation using mobile technologies: the potential mHealth approach. Front Psychol. 2014 Jun 10;5:559. doi: 10.3389/fpsyg.2014.00559. eCollection 2014. PMID 24959157
- [Background] Castelnuovo G, Zoppis I, Santoro E, Ceccarini M, Pietrabissa G, Manzoni GM, Corti S, Borrello M, Giusti EM, Cattivelli R, Melesi A, Mauri G, Molinari E, Sicurello F. Managing chronic pathologies with a stepped mHealth-based approach in clinical psychology and medicine. Front Psychol. 2015 Apr 14;6:407. doi: 10.3389/fpsyg.2015.00407. eCollection 2015. PMID 25926801
- [Background] Castelnuovo G, Manzoni GM, Villa V, Cesa GL, Pietrabissa G, Molinari E. The STRATOB study: design of a randomized controlled clinical trial of Cognitive Behavioral Therapy and Brief Strategic Therapy with telecare in patients with obesity and binge-eating disorder referred to residential nutritional rehabilitation. Trials. 2011 May 9;12:114. doi: 10.1186/1745-6215-12-114. PMID 21554734
- [Background] Cawley J, Meyerhoefer C, Biener A, Hammer M, Wintfeld N. Savings in Medical Expenditures Associated with Reductions in Body Mass Index Among US Adults with Obesity, by Diabetes Status. Pharmacoeconomics. 2015 Jul;33(7):707-22. doi: 10.1007/s40273-014-0230-2. PMID 25381647
- [Background] Cesa GL, Manzoni GM, Bacchetta M, Castelnuovo G, Conti S, Gaggioli A, Mantovani F, Molinari E, Cardenas-Lopez G, Riva G. Virtual reality for enhancing the cognitive behavioral treatment of obesity with binge eating disorder: randomized controlled study with one-year follow-up. J Med Internet Res. 2013 Jun 12;15(6):e113. doi: 10.2196/jmir.2441. PMID 23759286
- [Background] Cooper Z, Doll HA, Hawker DM, Byrne S, Bonner G, Eeley E, O'Connor ME, Fairburn CG. Testing a new cognitive behavioural treatment for obesity: A randomized controlled trial with three-year follow-up. Behav Res Ther. 2010 Aug;48(8):706-13. doi: 10.1016/j.brat.2010.03.008. PMID 20691328
- [Background] Deitel M. The International Obesity Task Force and "globesity". Obes Surg. 2002 Oct;12(5):613-4. doi: 10.1381/096089202321019558. No abstract available. PMID 12448379
- [Background] Epstein LH, Lin H, Carr KA, Fletcher KD. Food reinforcement and obesity. Psychological moderators. Appetite. 2012 Feb;58(1):157-62. doi: 10.1016/j.appet.2011.09.025. Epub 2011 Oct 8. PMID 22005184
- [Background] Ferron J, Ware W. Using randomization tests with responsive single-case designs. Behav Res Ther. 1994 Sep;32(7):787-91. doi: 10.1016/0005-7967(94)90037-x. PMID 7980366
- [Background] Fisher WW, Kelley ME, Lomas JE. Visual aids and structured criteria for improving visual inspection and interpretation of single-case designs. J Appl Behav Anal. 2003 Fall;36(3):387-406. doi: 10.1901/jaba.2003.36-387. PMID 14596583
- [Background] Forman EM, Hoffman KL, Juarascio AS, Butryn ML, Herbert JD. Comparison of acceptance-based and standard cognitive-based coping strategies for craving sweets in overweight and obese women. Eat Behav. 2013 Jan;14(1):64-8. doi: 10.1016/j.eatbeh.2012.10.016. Epub 2012 Nov 15. PMID 23265404
- [Background] Garcia-Garcia I, Horstmann A, Jurado MA, Garolera M, Chaudhry SJ, Margulies DS, Villringer A, Neumann J. Reward processing in obesity, substance addiction and non-substance addiction. Obes Rev. 2014 Nov;15(11):853-69. doi: 10.1111/obr.12221. Epub 2014 Sep 29. PMID 25263466
- [Background] Gifford EV, Lillis J. Avoidance and inflexibility as a common clinical pathway in obesity and smoking treatment. J Health Psychol. 2009 Oct;14(7):992-6. doi: 10.1177/1359105309342304. PMID 19786525
- [Background] Hayes S, Hogan M, Dowd H, Doherty E, O'Higgins S, Nic Gabhainn S, MacNeela P, Murphy AW, Kropmans T, O'Neill C, Newell J, McGuire BE. Comparing the clinical-effectiveness and cost-effectiveness of an internet-delivered Acceptance and Commitment Therapy (ACT) intervention with a waiting list control among adults with chronic pain: study protocol for a randomised controlled trial. BMJ Open. 2014 Jul 2;4(7):e005092. doi: 10.1136/bmjopen-2014-005092. PMID 24993763
- [Background] Howick J, Glasziou P, Aronson JK. The evolution of evidence hierarchies: what can Bradford Hill's 'guidelines for causation' contribute? J R Soc Med. 2009 May;102(5):186-94. doi: 10.1258/jrsm.2009.090020. No abstract available. PMID 19417051
- [Background] Kashdan TB, Barrios V, Forsyth JP, Steger MF. Experiential avoidance as a generalized psychological vulnerability: comparisons with coping and emotion regulation strategies. Behav Res Ther. 2006 Sep;44(9):1301-20. doi: 10.1016/j.brat.2005.10.003. PMID 16321362
- [Background] Lehnert T, Streltchenia P, Konnopka A, Riedel-Heller SG, Konig HH. Health burden and costs of obesity and overweight in Germany: an update. Eur J Health Econ. 2015 Dec;16(9):957-67. doi: 10.1007/s10198-014-0645-x. Epub 2014 Nov 8. PMID 25381038
- [Background] Lifshitz F, Lifshitz JZ. Globesity: the root causes of the obesity epidemic in the USA and now worldwide. Pediatr Endocrinol Rev. 2014 Sep;12(1):17-34. PMID 25345082
- [Background] Lillis J, Hayes SC, Bunting K, Masuda A. Teaching acceptance and mindfulness to improve the lives of the obese: a preliminary test of a theoretical model. Ann Behav Med. 2009 Feb;37(1):58-69. doi: 10.1007/s12160-009-9083-x. Epub 2009 Feb 28. PMID 19252962
- [Background] Manzoni GM, Pagnini F, Corti S, Molinari E, Castelnuovo G. Internet-based behavioral interventions for obesity: an updated systematic review. Clin Pract Epidemiol Ment Health. 2011 Mar 4;7:19-28. doi: 10.2174/1745017901107010019. PMID 21552423
- [Background] McCracken LM, Jones R. Treatment for chronic pain for adults in the seventh and eighth decades of life: a preliminary study of Acceptance and Commitment Therapy (ACT). Pain Med. 2012 Jul;13(7):860-7. doi: 10.1111/j.1526-4637.2012.01407.x. Epub 2012 Jun 8. PMID 22680627
- [Background] Pietrabissa G, Manzoni GM, Corti S, Vegliante N, Molinari E, Castelnuovo G. Addressing motivation in globesity treatment: a new challenge for clinical psychology. Front Psychol. 2012 Sep 3;3:317. doi: 10.3389/fpsyg.2012.00317. eCollection 2012. No abstract available. PMID 22969744
- [Background] Rachlin H. Free will from the viewpoint of teleological behaviorism. Behav Sci Law. 2007;25(2):235-50. doi: 10.1002/bsl.746. PMID 17393402
- [Background] Schuck K, Otten R, Kleinjan M, Bricker JB, Engels RC. Self-efficacy and acceptance of cravings to smoke underlie the effectiveness of quitline counseling for smoking cessation. Drug Alcohol Depend. 2014 Sep 1;142:269-76. doi: 10.1016/j.drugalcdep.2014.06.033. Epub 2014 Jul 5. PMID 25042212
- [Background] Thomas JJ, Koh KA, Eddy KT, Hartmann AS, Murray HB, Gorman MJ, Sogg S, Becker AE. Do DSM-5 eating disorder criteria overpathologize normative eating patterns among individuals with obesity? J Obes. 2014;2014:320803. doi: 10.1155/2014/320803. Epub 2014 Jun 26. PMID 25057413
- [Background] Tosolin F. Behavior-based safety. G Ital Med Lav Ergon. 2010 Jan-Mar;32(1 Suppl A):A7-12. No abstract available. English, Italian. PMID 20518200
- [Derived] Cattivelli R, Castelnuovo G, Musetti A, Varallo G, Spatola CAM, Riboni FV, Usubini AG, Tosolin F, Manzoni GM, Capodaglio P, Rossi A, Pietrabissa G, Molinari E. ACTonHEALTH study protocol: promoting psychological flexibility with activity tracker and mHealth tools to foster healthful lifestyle for obesity and other chronic health conditions. Trials. 2018 Nov 29;19(1):659. doi: 10.1186/s13063-018-2968-x. PMID 30486868